CLINICAL TRIAL: NCT01002794
Title: The Effect of Arthroscopic Partial Meniscectomy or Exercise Therapy as Treatment of Degenerative Meniscus Tears in Middle-aged Patients. A Randomized, Controlled Trial
Brief Title: Surgical or Exercise Therapy on Patients With Degenerative Meniscus Tears
Acronym: OMEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Southern Denmark (Other); South-Eastern Norway Regional Health Authority (Other)
Responsible Party: Principal Investigator, May Arna Risberg, Professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NARSDU2009
Record Dates: First submitted 2009-10-25; First posted 2009-10-27 (Estimated); Results first posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-02

CONDITIONS: Degenerative Meniscal Tear
Keywords: Degenerative meniscal tear; Arthroscopy; Exercise therapy
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Arthroscopic partial meniscectomy (Experimental): Standard arthroscopic partial meniscectomy - NGD 1
  Interventions: Procedure: Arthroscopic partial menisectomy
- Exercise Therapy (Experimental): Supervised neuromuscular- and strength training
  Interventions: Other: Supervised neuromuscular and strength training

INTERVENTIONS:
Procedure: Arthroscopic partial menisectomy — Standard arthroscopic partial meniscectomy, NGD 1. Carried out at Ullevaal University Hospital and Martina Hansens Hospital.
  Arms: Arthroscopic partial meniscectomy
Other: Supervised neuromuscular and strength training — Supervised exercise therapy in 12 weeks, both neuromuscular- and strength training. Carried out at Nimi Ullevaal Oslo or Gnist trending- og fysioterapi, Baerum
  Arms: Exercise Therapy

SUMMARY:
This study is conducted as a collaboration between NAR, Orthopedic Department, Oslo University Hospital,Ullevaal, Hjelp24Nimi Oslo, Martina Hansens Hospital Norway, and University of Southern Denmark, Odense, Denmark.

The investigators hypothesize that exercise is more effective than arthroscopic partial meniscectomy: a) on self-reported outcomes, functional performance and muscle strength in middle-aged patients subsequent to arthroscopic partial meniscectomy for a degenerative meniscus tear, and b) in preventing further development of knee osteoarthritis (OA).

DETAILED DESCRIPTION:
The aims of the study are:

1. At 3 months, to investigate the effect of arthroscopic partial meniscectomy versus exercise therapy on muscle strength and knee function in middle-aged patients with degenerative meniscus lesions.
2. At 2 years, to investigate the effect of arthroscopic partial meniscectomy versus exercise therapy on self-reported outcomes in middle aged patients with degenerative meniscus lesions.
3. At 5 years, to describe radiographic changes in knee osteoarthritis development after arthroscopic partial meniscectomy or exercise therapy in middle-aged patients with degenerative meniscus lesions.
4. 4. At 10 years, to describe radiographic changes in knee osteoarthritis development after arthroscopic partial meniscectomy or exercise therapy in middle-aged patients with degenerative meniscus lesions.

Patients included in the study will be randomized into one of two groups. The interventions are: arthroscopic partial meniscectomy and supervised neuromuscular- and strength training. Subjects will be tested before and after intervention, at 12 months, 24 months, five and 10 years.

Long-term follow-up studies are particularly important for this patient population. Both meniscal tears and partial meniscectomy has been demonstrated as risk factors for incident knee osteoarthritis and progression. However, it is not known whether the increased risk is due to the meniscal tear per se or resection of the meniscus. Furthermore, patients presenting with symptomatic degenerative meniscal tears have reduced knee muscle strength, which may be an additional risk factor for knee osteoarthritis. While knee muscle weakness has been shown to persist following surgery, the knowledge of long-term changes following surgical and non-surgical interventions for degenerative meniscal tears is limited. Accordingly, long-term between-group differences in muscle strength changes (at 5 and 10 years) and radiographic knee osteoarthritis changes (10 years) will also be investigated

ELIGIBILITY:
Inclusion Criteria:

* Age 35-60 years
* Knee pain for more than 2 months without a significant trauma
* Medial meniscal tear on MRI
* Eligible for arthroscopic partial meniscectomy
* Grade 0-2 radiographic severity (specification after Kellgren Lawrence)

Exclusion Criteria:

* Those requiring acute trauma surgeries, including those treated as acute cases in the ER
* Ligament injuries
* Tumours (MRI)
* Pain or other musculoskeletal comorbidities severely affecting lower extremity muscle function overriding the symptoms from the knee
* Grade 3 or 4 radiographic severity (specification after Kellgren Lawrence)
* Comorbidities excluding physical activities and exercise.
* Previous knee surgery within two years
* Not able to speak or read Norwegian, drug abuse or mental problems

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2024-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: May Arna Risberg, PT, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Orthopaedic Department, Oslo University Hospital, Ullevaal, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stensrud S, Risberg MA, Roos EM. Effect of exercise therapy compared with arthroscopic surgery on knee muscle strength and functional performance in middle-aged patients with degenerative meniscus tears: a 3-mo follow-up of a randomized controlled trial. Am J Phys Med Rehabil. 2015 Jun;94(6):460-73. doi: 10.1097/PHM.0000000000000209. PMID 25299520
- [Background] Kise NJ, Roos EM, Stensrud S, Engebretsen L, Risberg MA. The 6-m timed hop test is a prognostic factor for outcomes in patients with meniscal tears treated with exercise therapy or arthroscopic partial meniscectomy: a secondary, exploratory analysis of the Odense-Oslo meniscectomy versus exercise (OMEX) trial. Knee Surg Sports Traumatol Arthrosc. 2019 Aug;27(8):2478-2487. doi: 10.1007/s00167-018-5241-7. Epub 2018 Nov 16. PMID 30446783
- [Background] Kise NJ, Aga C, Engebretsen L, Roos EM, Tariq R, Risberg MA. Complex Tears, Extrusion, and Larger Excision Are Prognostic Factors for Worse Outcomes 1 and 2 Years After Arthroscopic Partial Meniscectomy for Degenerative Meniscal Tears: A Secondary Explorative Study of the Surgically Treated Group From the Odense-Oslo Meniscectomy Versus Exercise (OMEX) Trial. Am J Sports Med. 2019 Aug;47(10):2402-2411. doi: 10.1177/0363546519858602. Epub 2019 Jul 12. PMID 31298923
- [Background] Berg B, Roos EM, Kise NJ, Engebretsen L, Holm I, Risberg MA. On a Trajectory for Success-9 in Every 10 People With a Degenerative Meniscus Tear Have Improved Knee Function Within 2 Years After Treatment: A Secondary Exploratory Analysis of a Randomized Controlled Trial. J Orthop Sports Phys Ther. 2021 Jun;51(6):289-297. doi: 10.2519/jospt.2021.10025. Epub 2021 May 10. PMID 33971735
- [Result] Kise NJ, Risberg MA, Stensrud S, Ranstam J, Engebretsen L, Roos EM. Exercise therapy versus arthroscopic partial meniscectomy for degenerative meniscal tear in middle aged patients: randomised controlled trial with two year follow-up. BMJ. 2016 Jul 20;354:i3740. doi: 10.1136/bmj.i3740. PMID 27440192
- [Result] Berg B, Roos EM, Englund M, Kise NJ, Tiulpin A, Saarakkala S, Engebretsen L, Eftang CN, Holm I, Risberg MA. Development of osteoarthritis in patients with degenerative meniscal tears treated with exercise therapy or surgery: a randomized controlled trial. Osteoarthritis Cartilage. 2020 Jul;28(7):897-906. doi: 10.1016/j.joca.2020.01.020. Epub 2020 Mar 14. PMID 32184135
- [Result] Berg B, Roos EM, Kise NJ, Engebretsen L, Holm I, Risberg MA. Muscle Strength and Osteoarthritis Progression After Surgery or Exercise for Degenerative Meniscal Tears: Secondary Analyses of a Randomized Trial. Arthritis Care Res (Hoboken). 2022 Jan;74(1):70-78. doi: 10.1002/acr.24736. PMID 34151533
- [Derived] Berg B, Roos EM, Englund M, Kise NJ, Engebretsen L, Eftang CN, Risberg MA. Arthroscopic partial meniscectomy versus exercise therapy for degenerative meniscal tears: 10-year follow-up of the OMEX randomised controlled trial. Br J Sports Med. 2025 Jan 2;59(2):91-98. doi: 10.1136/bjsports-2024-108644. PMID 39326908
- [Derived] Kise NJ, Risberg MA, Stensrud S, Ranstam J, Engebretsen L, Roos EM. Exercise therapy versus arthroscopic partial meniscectomy for degenerative meniscal tear in middle aged patients: randomised controlled trial with two year follow-up. Br J Sports Med. 2016 Dec;50(23):1473-1480. doi: 10.1136/bjsports-2016-i3740rep. PMID 30142084
- [Derived] Stensrud S, Roos EM, Risberg MA. A 12-week exercise therapy program in middle-aged patients with degenerative meniscus tears: a case series with 1-year follow-up. J Orthop Sports Phys Ther. 2012 Nov;42(11):919-31. doi: 10.2519/jospt.2012.4165. Epub 2012 Sep 5. PMID 22960783

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arthroscopic Partial Meniscectomy | Exercise Therapy
Started | 70 | 70
Three Months | 60 | 63
One Year | 61 | 59
Two Years | 64 | 62
Five Years | 62 | 58
Completed | 62 | 58
Not Completed | 8 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arthroscopic Partial Meniscectomy | Exercise Therapy | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 70 | 70 | 140
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 48.9 [35 to 60] | 50.2 [35 to 60] | 49.6 [35 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 27 | 54
  Male | 43 | 43 | 86
Region of Enrollment [Number; unit: participants]
  Norway | 70 | 70 | 140

OUTCOME MEASURES:

1. Primary Outcome: KOOS4 - Change From Baseline
Description: The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a patient administered questionnaire containing 42 questions in 5 subscales concerning patient´s knee related pain, other knee symptoms, activity of daily life, sport and recreation and quality of life.Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
  KOOS4 is a composite score of the mean values of four of the five KOOS subscales (KOOS Pain, KOOS Symptoms, KOOS Sport/Rec and KOOS QOL).
Time Frame: 24 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arthroscopic Partial Meniscectomy | Exercise Therapy
Number analyzed (Participants) | 64 | 62
units on a scale | 24.4 [20.7 to 28.0] | 25.3 [21.6 to 29.0]
Statistical Analysis 1: Comparison: Arthroscopic Partial Meniscectomy vs Exercise Therapy; Power calculation: The sample size calculation was based on the change in KOOS4 from baseline to two year follow-up. To detect a 10 point difference with a standard deviation of 15, with a level of power of 90%, level of significance of 0.05, and an estimated 15% dropout rate at two years, we determined that we would need 56 participants in each group. To allow for a 20% crossover rate, we randomised 140 participants; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis

2. Primary Outcome: Peak Torque Knee Extension - Change From Baseline
Description: Peak torque knee extension (Newton meter) - Change from baseline
Time Frame: at 3 months
Measure: Mean (95% Confidence Interval); unit: Newton meter
Arm/Group | Arthroscopic Partial Meniscectomy | Exercise Therapy
Number analyzed (Participants) | 60 | 63
Newton meter | -2.63 [-8.7 to 3.4] | 20.7 [14.7 to 26.7]

3. Primary Outcome: Peak Torque Knee Flexion - Change From Baseline
Description: Peak torque knee flexion (Newton meter) - Change from baseline
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: Newton meter
Arm/Group | Arthroscopic Partial Meniscectomy | Exercise Therapy
Number analyzed (Participants) | 60 | 63
Newton meter | 5.0 [1.6 to 8.4] | 12.8 [9.4 to 16.2]

4. Primary Outcome: Knee Osteoarthritis Incidence
Description: In line with baseline assessment of the tibiofemoral joint, standing radiographs of the tibiofemoral joint is taken bilaterally with a Synaflexer Frame (Synarc Inc) that ensure alignment of the x-ray beam and standardize the placement of the knee in approximately 20 degrees of flexion and 5 degrees of external rotation for an anterior-posterior view. A sagittal view is also taken with the knee in flexion. Kellgren and Lawrence will be used for classification in addition to description of osteophytes and joint Space narrowing (JSN) will be measured.
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arthroscopic Partial Meniscectomy | Exercise Therapy
Number analyzed (Participants) | 62 | 58
Participants | 10 | 9

5. Primary Outcome: Radiographic Progression (the Osteoarthritis Research Society International [OARSI] Atlas) [Time Frame: At 10 Years]
Description: Radiographic progression based on the sum of marginal tibiofemoral osteophyte grades and tibiofemoral joint space narrowing (the Osteoarthritis Research Society International [OARSI] atlas) [Time Frame: At 10 years]
Time Frame: 10 years
Reporting Status: Not Posted, anticipated posting 2024-12

6. Secondary Outcome: One Leg Hop Test - Change From Baseline
Description: Change in distance (meters) hopped on the One leg hop test from baseline to three months (higher is better).
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: Meters
Arm/Group | Arthroscopic Partial Meniscectomy | Exercise Therapy
Number analyzed (Participants) | 60 | 63
Meters | 6.1 [1.4 to 10.8] | 11.0 [6.4 to 15.7]

7. Secondary Outcome: 6 Meter Timed Hop Test - Change From Baseline
Description: Change in time (seconds) on the 6 meter timed hop test from baseline to 3 months (lower is better)
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: Seconds
Arm/Group | Arthroscopic Partial Meniscectomy | Exercise Therapy
Number analyzed (Participants) | 60 | 63
Seconds | -0.1 [-0.4 to 0.1] | -0.5 [-0.8 to -0.3]

8. Secondary Outcome: Knee Bends 30 Sec - Change From Baseline
Description: Change in number of repetitions performed on the Knee bends 30 seconds test from baseline to 3 months (higher is better).
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: Number of repetitions
Arm/Group | Arthroscopic Partial Meniscectomy | Exercise Therapy
Number analyzed (Participants) | 60 | 63
Number of repetitions | 8.5 [6.6 to 10.4] | 9.9 [8.1 to 11.8]

9. Secondary Outcome: Peak Torque Knee Extension - Change From Baseline
Description: Change in Peak torque knee extension (Newton meter) from baseline to 12 months (higher is better).
Time Frame: 1 year
Measure: Mean (95% Confidence Interval); unit: Newton meter
Arm/Group | Arthroscopic Partial Meniscectomy | Exercise Therapy
Number analyzed (Participants) | 61 | 59
Newton meter | 8.8 [2.8 to 14.8] | 18.2 [12.1 to 24.4]

10. Secondary Outcome: Peak Torque Knee Flexion - Change From Baseline
Description: Change in Peak torque knee flexion (Newton meter) from baseline to 12 months (higher is better).
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: Netwon meter
Arm/Group | Arthroscopic Partial Meniscectomy | Exercise Therapy
Number analyzed (Participants) | 61 | 59
Netwon meter | 4.3 [0.9 to 7.7] | 11.4 [7.9 to 14.8]

11. Secondary Outcome: One-leg Hop Test - Change in From Baseline
Description: Change in distance (meters) hopped on the One leg hop test from baseline to 12 months (higher is better).
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: Meters
Arm/Group | Arthroscopic Partial Meniscectomy | Exercise Therapy
Number analyzed (Participants) | 61 | 59
Meters | 13.1 [8.3 to 17.8] | 13.2 [8.4 to 17.9]

12. Secondary Outcome: 6 Meter Timed Hop Test - Change From Baseline
Description: Change in time (seconds) on the 6 meter timed hop test from baseline to 12 months (lower is better).
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: Seconds
Arm/Group | Arthroscopic Partial Meniscectomy | Exercise Therapy
Number analyzed (Participants) | 61 | 59
Seconds | -0.3 [-0.5 to -0.0] | -0.6 [-0.8 to -0.4]

13. Secondary Outcome: Knee Bends 30 Sec - Change From Baseline
Description: Change in number of repetitions performed on the Knee bends 30 seconds test from baseline to 12 months (higher is better).
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: Number of repetitions
Arm/Group | Arthroscopic Partial Meniscectomy | Exercise Therapy
Number analyzed (Participants) | 61 | 59
Number of repetitions | 10.6 [8.7 to 12.5] | 9.2 [7.3 to 11.1]

14. Secondary Outcome: KOOS Pain - Change From Baseline
Description: Change in the Knee Injury and Osteoarthritis Outcome Score (KOOS) Pain subscale from baseline to two years.
  Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
Time Frame: 24 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arthroscopic Partial Meniscectomy | Exercise Therapy
Number analyzed (Participants) | 64 | 62
units on a scale | 21.7 [18.0 to 25.5] | 23.2 [19.4 to 27.0]

15. Secondary Outcome: KOOS Symptoms - Change From Baseline
Description: Change in the Knee Injury and Osteoarthritis Outcome Score (KOOS) Symptoms subscale from baseline to two years. Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
Time Frame: 24 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arthroscopic Partial Meniscectomy | Exercise Therapy
Number analyzed (Participants) | 64 | 62
units on a scale | 12.0 [8.7 to 15.4] | 17.4 [14.0 to 20.9]

16. Secondary Outcome: KOOS ADL - Change From Baseline
Description: Change in the Knee Injury and Osteoarthritis Outcome Score (KOOS) Activities in Daily Living (ADL) subscale from baseline to two years.
  Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale
Time Frame: 24 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arthroscopic Partial Meniscectomy | Exercise Therapy
Number analyzed (Participants) | 64 | 62
units on a scale | 13.8 [10.7 to 16.9] | 15.4 [12.2 to 18.6]

17. Secondary Outcome: KOOS Sport/Rec - Change From Baseline
Description: Change in the Knee Injury and Osteoarthritis Outcome Score (KOOS) Sport and recreation (Sport/Rec) subscale from baseline to two years.
  Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
Time Frame: 24 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arthroscopic Partial Meniscectomy | Exercise Therapy
Number analyzed (Participants) | 64 | 62
units on a scale | 30.8 [25.4 to 36.1] | 29.3 [24.0 to 34.7]

18. Secondary Outcome: KOOS QOL - Change From Baseline
Description: Change in the Knee Injury and Osteoarthritis Outcome Score (KOOS) Quality of Life (QOL) subscale from baseline to two years.
  Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
Time Frame: 24 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arthroscopic Partial Meniscectomy | Exercise Therapy
Number analyzed (Participants) | 64 | 62
units on a scale | 33.1 [28.7 to 37.5] | 31.3 [26.8 to 35.7]

19. Secondary Outcome: SF-36 MCS - Change From Baseline
Description: Change in Short form 36 mental component summary (SF-36 MCS) from baseline to 24 months (range: 0-100; higher is better)
Time Frame: 24 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arthroscopic Partial Meniscectomy | Exercise Therapy
Number analyzed (Participants) | 64 | 62
units on a scale | -0.3 [-2.0 to 1.4] | 1.1 [-1.1 to 3.3]

20. Secondary Outcome: SF-36 PCS - Change From Baseline
Description: Change in Short form 36 physical component summary (SF-36 PCS) from baseline to 24 months (range: 0-100; higher is better)
Time Frame: 24 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arthroscopic Partial Meniscectomy | Exercise Therapy
Number analyzed (Participants) | 64 | 62
units on a scale | 7.0 [5.3 to 8.6] | 5.5 [3.5 to 7.4]

21. Secondary Outcome: KOOS Pain Subscale - Change From Baseline
Description: Change in the Knee Injury and Osteoarthritis Outcome Score (KOOS) Pain subscale from baseline to five years (range: 0-100; higher is better).
Time Frame: 5 years
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arthroscopic Partial Meniscectomy | Exercise Therapy
Number analyzed (Participants) | 62 | 57
units on a scale | 23.8 [20.1 to 27.5] | 21.3 [17.4 to 25.2]

22. Secondary Outcome: KOOS Symptoms Subscale - Change From Baseline
Description: Change in the Knee Injury and Osteoarthritis Outcome Score (KOOS) Symptoms subscale from baseline to five years (range: 0-100; higher is better).
Time Frame: 5 years
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arthroscopic Partial Meniscectomy | Exercise Therapy
Number analyzed (Participants) | 62 | 57
units on a scale | 12.9 [9.1 to 16.7] | 13.2 [9.3 to 17.2]

23. Secondary Outcome: KOOS ADL Subscale - Change From Baseline
Description: Change in the Knee Injury and Osteoarthritis Outcome Score (KOOS) Activities of Daily Living (ADL) subscale from baseline to five years (range: 0-100; higher is better).
Time Frame: 5 years
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arthroscopic Partial Meniscectomy | Exercise Therapy
Number analyzed (Participants) | 62 | 57
units on a scale | 14.5 [11.5 to 17.5] | 14.6 [11.5 to 17.8]

24. Secondary Outcome: KOOS Sport/Rec Subscale - Change From Baseline
Description: Change in the Knee Injury and Osteoarthritis Outcome Score (KOOS) Sport and Recreation (Sport/Rec) subscale from baseline to five years (range: 0-100; higher is better).
Time Frame: 5 years
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arthroscopic Partial Meniscectomy | Exercise Therapy
Number analyzed (Participants) | 62 | 57
units on a scale | 33.4 [27.5 to 39.3] | 29.0 [22.9 to 35.1]

25. Secondary Outcome: KOOS QOL Subscale - Change From Baseline
Description: Change in the Knee Injury and Osteoarthritis Outcome Score (KOOS) Quality of Life (QOL) subscale from baseline to five years (range: 0-100; higher is better).
Time Frame: 5 years
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arthroscopic Partial Meniscectomy | Exercise Therapy
Number analyzed (Participants) | 62 | 57
units on a scale | 34.4 [29.3 to 39.4] | 30.7 [25.5 to 36.0]

26. Secondary Outcome: Peak Torque Knee Extension - Change From Baseline
Description: Change in body weight (kilograms) normalized Peak torque knee extension (Newton meter/kg) from baseline to five years (higher is better).
Time Frame: 5 years
Measure: Mean (95% Confidence Interval); unit: Newton meters/kg
Arm/Group | Arthroscopic Partial Meniscectomy | Exercise Therapy
Number analyzed (Participants) | 59 | 57
Newton meters/kg | 0.03 [-0.05 to 0.10] | 0.13 [0.05 to 0.20]

27. Secondary Outcome: Peak Torque Knee Flexion - Change From Baseline
Description: as for outcome 26
Time Frame: 5 years
Measure: Mean (95% Confidence Interval); unit: Newton meters/kg
Arm/Group | Arthroscopic Partial Meniscectomy | Exercise Therapy
Number analyzed (Participants) | 59 | 57
Newton meters/kg | -0.02 [-0.07 to 0.02] | 0.04 [0.00 to 0.09]

28. Secondary Outcome: Knee Osteoarthritis Incidence (Kellgren and Lawrence Classification )
Description: Knee osteoarthritis incidence (Kellgren and Lawrence classification) [ Time Frame: 10 years]
Time Frame: 10 years
Reporting Status: Not Posted, anticipated posting 2024-12

29. Secondary Outcome: KOOS4 - Change From Baseline
Description: Change in KOOS4 from baseline to 10 years (range: 0-100; higher is better). KOOS4 is a composite score of the mean values of four of the five Knee Injury and Osteoarthritis Outcome Score (KOOS) subscales (KOOS Pain, KOOS Symptoms, KOOS Sport/Rec and KOOS QOL).
Time Frame: 10 years
Reporting Status: Not Posted, anticipated posting 2024-12

30. Secondary Outcome: KOOS Pain Subscale - Change From Baseline
Description: Change in the Knee Injury and Osteoarthritis Outcome Score (KOOS) Pain subscale from baseline to 10 years (range: 0-100; higher is better).
Time Frame: 10 years
Reporting Status: Not Posted

31. Secondary Outcome: KOOS Symptoms Subscale - Change From Baseline
Description: Change in the Knee Injury and Osteoarthritis Outcome Score (KOOS) Symptoms subscale from baseline to 10 years (range: 0-100; higher is better).
Time Frame: 10 years
Reporting Status: Not Posted, anticipated posting 2024-12

32. Secondary Outcome: KOOS ADL Subscale - Change From Baseline
Description: Change in the Knee Injury and Osteoarthritis Outcome Score (KOOS) Activities of Daily Living (ADL) subscale from baseline to 10 years (range: 0-100; higher is better).
Time Frame: 10 years
Reporting Status: Not Posted, anticipated posting 2024-12

33. Secondary Outcome: KOOS Sport/Rec Subscale - Change From Baseline
Description: as for outcome 24
Time Frame: 10 years
Reporting Status: Not Posted, anticipated posting 2024-12

34. Secondary Outcome: KOOS QOL Subscale - Change From Baseline
Description: Change in the Knee Injury and Osteoarthritis Outcome Score (KOOS) Quality of Life (QOL) subscale from baseline to ten years (range: 0-100; higher is better).
Time Frame: 10 years
Reporting Status: Not Posted, anticipated posting 2024-12

35. Secondary Outcome: Peak Torque Knee Flexion - Change From Baseline
Description: Change in body weight (kilograms) normalized Peak torque knee flexion (Newton meter/kg) from baseline to ten years (higher is better).
Time Frame: 10 years
Reporting Status: Not Posted, anticipated posting 2024-12

36. Secondary Outcome: Peak Torque Knee Extension - Change From Baseline
Description: Change in body weight (kilograms) normalized Peak torque knee extension (Newton meter/kg) from baseline to 10 years (higher is better).
Time Frame: 10 years
Reporting Status: Not Posted, anticipated posting 2024-12

ADVERSE EVENTS:
Groups:
- Arthroscopic Partial Meniscectomy: Standard arthroscopic partial meniscectomy - NGD 1
  Arthroscopic partial menisectomy: Standard arthroscopic partial meniscectomy, NGD 1. Carried out at Ullevaal University Hospital and Martina Hansens Hospital.
  Adverse events related to the surgical procedure; i.e. lung embolus, infection, acute heart attac.
- Exercise Therapy: Supervised neuromuscular- and strength training
  Supervised neuromuscular and strength training: Supervised exercise therapy in 12 weeks, both neuromuscular- and strength training. Carried out at Nimi Ullevaal Oslo or Gnist trending- og fysioterapi, Baerum
  Adverse events related to the exercise; i.e. heart- og lung disease, trauma
Arm/Group | Arthroscopic Partial Meniscectomy | Exercise Therapy
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/70
Other Adverse Events (participants affected / at risk) | 0/70 | 0/70

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No